CLINICAL TRIAL: NCT04931173
Title: Is Mechanical Bowel Preparation Necessary to Reduce Surgical Site Infection Following Colon Surgery: a Randomized Controlled Trial
Brief Title: Mechanical Bowel Prep Randomized Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Erin Kennedy, Colorectal Surgeon; Department Head, Division of General Surgery, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PJT-165836
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Surgery
Keywords: Surgical Site Infection; Mechanical Bowel Preparation; Randomized Controlled Trial
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, parallel, two-arm, non-inferiority randomized controlled trial comparing IVA+OA+MBP versus IVA+OA to reduce surgical site infection following colon surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: IV and Oral antibiotics (IVA+OA) (Active Comparator): Patients will receive cefazolin 2g IV and metronidazole 500 mg IV administered by the anesthesiologist within 60 minutes prior to the skin incision on the day of surgery. Standardized re-dosing of cefazolin 2g IV will occur every 4 hours and metronidazole 500 mg IV will occur every 8 hours during the surgical procedure. Following surgery, no further IVA will be given for SSI prophylaxis. In addition, patients will self-administer 1g neomycin and 1g metronidazole orally at 1500, 1700 and 2300 hours the day before surgery. Following this, they will not receive any further OAs for SSI prophylaxis.
  Interventions: Other: IVA+OA versus IVA+MBP+OA
- Group B: IV antibiotics, MBP and oral antibiotics (IVA+MBP+OA) (Active Comparator): Patients will receive IVA and OA per Group A. In addition, patients will stay on clear fluids and self-administer a 2L polyethylene glycol MBP orally, between 1500 and 2300 hours on the day before surgery.
  Interventions: Other: IVA+OA versus IVA+MBP+OA

INTERVENTIONS:
Other: IVA+OA versus IVA+MBP+OA — Non-inferiority RCT comparing IVA+OA+MBP vs IVA+OA to reduce surgical site infection following colon surgery

SUMMARY:
Following colon surgery, surgical site infection (SSI) is the most common complication and leads to longer recovery time for patients and increased health care costs. Currently, there is high quality evidence to show that the combination of intravenous antibiotics (IVA), mechanical bowel preparation (MBP) and oral antibiotics (OA) is the most effective bowel preparation to reduce SSI. However, there are no studies comparing IVA+MBP+OA and IVA+OA. This is an important question because if IVA+OA works the same as IVA+MBP+OA, then MBP may be safely omitted as part of the bowel preparation to reduce SSI and patients would avoid the side effects of MBP prior to their surgery. Therefore, the objective is to perform a trial to determine if IVA+OA works the same as IVA+MBP+OA to reduce SSI following colon surgery.

DETAILED DESCRIPTION:
Background: Colon surgery includes surgery for colon cancer, inflammatory bowel disease and other benign disease such as diverticulitis. In Canada, approximately 21,000 colon surgeries are performed annually. Following colon surgery, the most common complication is surgical site infection (SSI) and rates of up to 25% have been reported. The high volume of colon cancer surgery, coupled with high rates of SSI lead to considerably worse health care outcomes for patients including increased recovery time, length of stay and readmission. Currently, several different bowel preparations to reduce SSI are being used in Canada and there is significant practice variation due to lack of RCTs and conflicting practice guidelines. More recently, several large observational studies and a network meta-analysis have shown that a combination of intravenous antibiotics, mechanical bowel preparation and oral antibiotics (IVA+MBP+OA) is superior to IVA+MBP and IVA alone. Interestingly, these studies also showed that SSI rates for IVA+OA are comparable to IVA+MBP+OA. These data provide a strong rationale to conduct a RCT comparing IVA+OA versus IVA+MBP+OA to determine if MBP is a necessary part of the bowel preparation or if MBP can be safely omitted and the side effects of MBP avoided.

Objectives: Therefore, the objectives are to conduct a multi-centre, parallel, two arm, non-inferiority RCT comparing IVA+MBP+OA versus IVA+OA to reduce SSI following colon surgery.

Methods: The inclusion criteria are any patient (i) undergoing elective colon surgery, (ii) over the age of 18 years and (3) provides informed consent. Eligible patients at 4 centres across Canada will be randomized to one of two groups: IVA+OA+MBP or IVA+OA. The primary outcome for the trial is the overall rate of SSI at 30 days following surgery. Assuming an overall SSI rate of 7% with IVA+MBP+OA and a non-inferiority margin of 4.0%, 1062 patients will be required with a one sided alpha of 0.05 and a power of 80%. This non-inferiority margin was unanimously accepted as clinically meaningful by all of the Site Leads at participating centres. Primary analyses will be performed per-protocol in patients who received treatment as allocated and underwent colon surgery. Overall SSI rates at 30 days following surgery will be compared using a general linear model and non-inferiority will be declared if the upper limit of the one sided 95% confidence interval of the absolute risk difference of overall SSI following surgery does not include 4.0%.

Relevance: This trial will be highly relevant to both patients and physicians as the results will provide definitive, high quality, patient-centred evidence about whether MBP is a necessary part of the optimal bowel preparation to reduce SSI and improve both patient experience and outcomes. These results will have significant potential to change practice in Canada and world-wide.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective colon surgery for benign or malignant disease
* over the age of 18 years
* provides informed consent.

Exclusion Criteria:

* known anaphylaxis to neomycin or metronidazole
* pregnancy or lactation
* chronic renal failure (serum creatinine > 220 umol/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | 30 days following date of surgery
  Rate of overall surgical site infection

SECONDARY OUTCOMES:
Patient tolerability of the bowel preparation | 5 minutes (completed in pre-operative holding area on the day of surgery)
  Validated 9-item questionnaire entitled: "Mayo Clinic Bowel Prep Tolerability Questionnaire" (Scale 1-4; lower score = better outcome)
Length of stay | 2-7 days
  length of stay in hospital following colorectal procedure
30-day ER rate | 30 days
  emergency room visit rate to any hospital within 30 days of surgery
30-day readmission rate | 30 days
  readmission rate to any hospital within 30 days of surgery

REFERENCES:
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942